CLINICAL TRIAL: NCT01118260
Title: TIVA Versus Spinal Anaesthesia in Patients Undergoing Transurethral Prostate Resection
Brief Title: Total Intravenous Anaesthesia (TIVA) Versus Spinal Anaesthesia in Patients Undergoing Transurethral Prostate Resection
Acronym: TURPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Dr. med. Vegard Dahl, Asker & Baerum Hospital, Vestre Viken HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-002672-42
Record Dates: First submitted 2010-04-07; First posted 2010-05-06 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-05

CONDITIONS: Prostate; Hyperplasia
Keywords: prostata hyperplasia; transurethral resection; TIVA; spinal anaesthesia
MeSH Terms: conditions — Hyperplasia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIVA (Active Comparator): Total intravenous anaesthesia (TIVA) with propofol and remifentanil
  Interventions: Procedure: total intravenous anaesthesia
- Spinal (Active Comparator): Spinal anaesthesia with bupivacaine and fentanyl
  Interventions: Procedure: spinal anaesthesia

INTERVENTIONS:
Procedure: total intravenous anaesthesia — propofol and remifentanil
  Arms: TIVA
Procedure: spinal anaesthesia — bupivacaine and fentanyl
  Arms: Spinal

SUMMARY:
Comparison of total intravenous anaesthesia with spinal anaesthesia in patients undergoing transurethral prostate resection

DETAILED DESCRIPTION:
Comparison of total intravenous anaesthesia with spinal anaesthesia in patients undergoing transurethral prostate resection regarding patient satisfaction and discharge time

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* signed informed consent
* elective transurethral prostata resection

Exclusion Criteria:

* ASA more than 3
* kidney disease, liver disease
* intolerance against bupivacaine, fentanyl, propofol og remifentanil
* chronic pulmonary disease
* dementia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 4 hours
  Patient satisfaction was measured asking the patient about satisfaction with anaesthesia using a 5-point Linkert scale: totally satisfied - satisfied - neither satisfied nor dissatisfied - dissatisfied - totally dissatisfied Time frame: Start anaesthesia to end post anaesthestic care unit

SECONDARY OUTCOMES:
time in PACU | 4 hours
  period in post anaesthetic care unit

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Dahl, MD, PhD, Study Chair — Asker & Baerum Hospital; Elisabet Andersson, Principal Investigator — Asker & Baerum Hospital
Locations (1):
- Asker & Baerum Hospital, Rud, Norway